CLINICAL TRIAL: NCT00161382
Title: HIV Prevention Programs for Middle School Students
Brief Title: Development and Evaluation of an HIV, STD, and Pregnancy Prevention Program for Middle School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Tortolero, ◦Allan King Professorship in Public Health & Director, Center for Health Promotion and Prevention Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH066640 (NIH); R01MH066640-01 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Pregnancy
Keywords: HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): HIV, STD, and pregnancy prevention curriculum
  Interventions: Behavioral: HIV, STD, and pregnancy prevention curriculum
- Control Group (Experimental): Standard sexual education curriculum
  Interventions: Behavioral: Standard sexual education curriculum

INTERVENTIONS:
Behavioral: HIV, STD, and pregnancy prevention curriculum — This HIV, STD, and pregnancy intervention program entitled, "It's Your Game...Keep it Real", consists of 12 lessons delivered in Grades 7 and 8. In each grade, the program integrates group-based classroom activities (e.g., role plays, group discussion, small group activities) with personalized journaling and individual tailored activities delivered on laptop computers. A life skills decision-making paradigm (Select, Detect, Protect) underlies the activities, teaching students to select personal limits regarding risk behaviors, to detect signs or situations that might challenge these limits, and to use refusal skills and other tactics to protect these limits.
  Arms: Intervention Group
Behavioral: Standard sexual education curriculum — Control curriculum consists of standard sexual education.
  Arms: Control Group

SUMMARY:
This study will develop and evaluate a school-based HIV, STD, and pregnancy prevention program for 7th and 8th grade middle school students.

DETAILED DESCRIPTION:
The purpose of this study is to develop and evaluate a school-based HIV, STD, and pregnancy prevention program for 7th and 8th grade middle school students using a randomized-controlled intervention trial. The intervention program consists of a classroom-based curriculum and an interactive CD-ROM. Ten middle schools were recruited to participate in this intervention trial. Five middle schools were randomized to the intervention group; and five middle schools were randomized to the control group. The study is also developing a model for obtaining community support for the development of HIV, STD and pregnancy prevention programs for middle school youth.

The primary hypothesis to be tested is: Students attending middle schools who receive a multi-component HIV, STD, pregnancy prevention intervention will postpone sexual activity or reduce levels of current sexual activity relative to those in the comparison condition. The major dependent variables are proportion of students that are sexually active, and the proportion initiating sexual intercourse. Intentions to engage in sexual activity, number of times of unprotected sexual intercourse, and number of sexual partners will also be examined. Secondary hypotheses will examine the effect of the multi-component HIV, STD, and pregnancy prevention intervention on the student's knowledge, self-efficacy, attitudes, perceived norms, barriers, and communication with parents.

The specific aims of this project are to:

1. Develop a model for obtaining community-based support for HIV, STD, and pregnancy prevention interventions for middle school students.
2. Adapt a tested, school-based, HIV, STD, and pregnancy prevention curriculum for middle school students using qualitative data from the target population, parents, and community representatives.
3. Develop an interactive CD-ROM-based tailored HIV, STD and pregnancy prevention intervention to provide individualized learning opportunities for middle school students.
4. Evaluate the effect of the multi-component intervention (classroom curriculum and CD-ROM intervention) on sexual behavior outcomes (proportion of students who initiate sexual intercourse, proportion of currently sexually active students having unprotected sexual intercourse, number of sexual partners, and intentions to have sexual intercourse) among middle school students.
5. Evaluate the effect of the multi-component intervention on student impact variables such as knowledge, self-efficacy, attitudes, barriers, and perceived norms related to sexual risk-taking behavior and academic achievement among middle school students.
6. Disseminate findings to the scientific community, school districts, and community agencies.

ELIGIBILITY:
Inclusion Criteria:

* 7th Grade
* Attend one of the ten recruited schools

Exclusion Criteria:

* Non-English speaking
* Physical disability that prevents student from completing intervention and survey

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3007 (Actual)
Dates: Start 2002-09; Primary Completion 2007-03 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R. Tortolero, PhD, Principal Investigator — University of Texas Houston Health Science Center - School of Public Health; Christine M. Markham, PhD, Principal Investigator — University of Texas Houston Health Science Center - School of Public Health
Locations (1):
- University of Texas Houston Health Science Center - School of Public Health, Houston, Texas, United States

REFERENCES:
- [Result] Tortolero SR, Markham CM, Peskin MF, Shegog R, Addy RC, Escobar-Chaves SL, Baumler ER. It's Your Game: Keep It Real: delaying sexual behavior with an effective middle school program. J Adolesc Health. 2010 Feb;46(2):169-79. doi: 10.1016/j.jadohealth.2009.06.008. Epub 2009 Aug 18. PMID 20113923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 3,007 participants who were recruited for the study, 371 were excluded because of limited English proficiency and 1,191 were excluded because they did not obtain parental affirmative consent. Thus, 1,445 participants were randomized to either the comparison (n = 847) or the intervention (n = 598) condition.
Groups:
- Intervention Group: Participants receiving HIV, STD, and pregnancy prevention curriculum
  HIV, STD, Pregnancy Prevention Curriculum: This HIV, STD, and pregnancy intervention program entitled, "It's Your Game...Keep it Real", consists of 12 lessons delivered in Grades 7 and 8. In each grade, the program integrates group-based classroom activities (e.g., role plays, group discussion, small group activities) with personalized journaling and individual tailored activities delivered on laptop computers. A life skills decision-making paradigm (Select, Detect, Protect) underlies the activities, teaching students to select personal limits regarding risk behaviors, to detect signs or situations that might challenge these limits, and to use refusal skills and other tactics to protect these limits.
- Control Group: No intervention: Control curriculum consists of standard sexual education.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 598 (Number of students allocated to intervention group) | 847 (Number of students allocated to comparison group)
Completed | 349 (Number of intervention students included in the analyzed cohort (i.e., completed 9th-grade survey)) | 558 (Number of control students included in the analyzed cohort (i.e., completed 9th-grade survey))
Not Completed | 249 | 289

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 349 | 558 | 907
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (.57) | 13.0 (.51) | 13.0 (.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 326 | 536
  Male | 139 | 232 | 371

OUTCOME MEASURES:

1. Primary Outcome: Initiation of Sexual Intercourse
Description: The effect of the intervention on delayed sexual initiation at the 9th-grade follow-up for those students who reported no lifetime sexual activity at baseline was assessed as the primary outcome. The primary hypothesis tested was that the intervention would decrease the number of adolescents who initiated sexual activity by the ninth grade relative to those in the comparison schools. Sexual activity was defined as participation in vaginal, oral, or anal sex. Sexual activity questions were defined in advance and were worded in a gender-neutral manner to illicit responses for same and opposite-sex partners.
Time Frame: Measured throughout the study, and at 2006/2007 school year
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 349 | 558
participants | 308 | 509

2. Secondary Outcome: Knowledge
Time Frame: Measured throughout the study
Reporting Status: Not Posted

3. Secondary Outcome: Self-efficacy
Time Frame: Measured throughout the study
Reporting Status: Not Posted

4. Secondary Outcome: Attitudes
Time Frame: Measured throughout the study
Reporting Status: Not Posted

5. Secondary Outcome: Perceived Norms
Time Frame: Measured throughout the study
Reporting Status: Not Posted

6. Secondary Outcome: Barriers
Time Frame: Measured throughout the study
Reporting Status: Not Posted

7. Secondary Outcome: Communication With Parents
Time Frame: Measured throughout the study
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Students That Are Sexually Active
Time Frame: Measured over a period of 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and Other [Non-Serious] Adverse Events were not collected/assessed
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No